CLINICAL TRIAL: NCT07320248
Title: Evaluating the Efficacy of Virtual Reality in Patient Preparation for Cardiac Catheterization Procedures in Oman: A Randomized Controlled Trial
Brief Title: Virtual Reality for Patient Preparation Before Cardiac Catheterization in Oman
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 107/2025
Record Dates: First submitted 2025-09-13; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease; Ischaemic Heart Desease; Cardiac Catheterization
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants and care providers will be aware of group allocation due to the nature of the intervention. However, the outcomes assessor analyzing the questionnaire data will be blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Pre-procedure Education (Experimental): Participants in this group will receive a virtual reality-based educational session prior to their first cardiac catheterization. The VR module will provide a 3D immersive orientation to the catheterization process, including admission, preparation, transfer to the Cath Lab, procedural steps, and post-procedure recovery. The VR experience will last approximately 10-15 minutes and will be delivered once in a quiet setting within the hospital prior to the scheduled procedure. This innovative approach aims to reduce anxiety and enhance understanding of the procedure, ultimately improving patient outcomes. By familiarizing participants with the environment and steps involved, the program seeks to empower them and give them control over their healthcare experience.
  Interventions: Behavioral: Virtual Reality Education
- Standard Pre-procedure Education (No Intervention): Participants in this group will receive the usual standard education provided at the hospital, which includes a verbal explanation by the nurse or physician and a written patient information leaflet describing the procedure, expected preparation, and recovery process. The session will last approximately 10-15 minutes and will be conducted prior to the scheduled procedure. During this time, participants will have the opportunity to ask questions and clarify any concerns they may have regarding their treatment. This interactive approach aims to enhance understanding and ensure that everyone feels confident and informed before proceeding.

INTERVENTIONS:
Behavioral: Virtual Reality Education — Participants in this group will receive a virtual reality-based educational session prior to their first cardiac catheterization. The VR module provides an immersive 3D orientation to the catheterization process, including admission, preparation, transfer to the Cath Lab, procedural steps, and post-procedure recovery. The VR session lasts approximately 10-15 minutes and is delivered once in a quiet hospital setting before the scheduled procedure. This innovative approach aims to enhance patient understanding and reduce anxiety associated with the catheterization experience. By familiarizing participants with the entire process beforehand, the program seeks to improve overall satisfaction and outcomes.
  Arms: Virtual Reality Pre-procedure Education

SUMMARY:
Background: Cardiovascular disease is considered one of the most prevalent diseases in recent times, and cardiac catheterization is widely used to diagnose and treat cardiovascular disease. However, patients often experience significant anxiety before the procedure due to fear of the unknown, potential complications, and concern about discomfort.Aim: To evaluate the efficacy of virtual reality technology to reduce anxiety and improve patient satisfaction, attitude, and usefulness in individuals undergoing first-time cardiac catheterization procedures in Oman.Method: A mixed-method randomized control trial will be used with approximately 120 patients from different tertiary hospitals in Oman. The experimental group will experience a virtual reality simulation of the catheterization process before providing informed consent, while the control group will receive the standard pre-procedure education. The Arabic version of the DASS-21 scale will be used to assess anxiety level pre- and post-intervention, while patient satisfaction will be measured through qualitative interviews with a subset of 10 participants.Result: ANOVA will be conducted to examine differences in anxiety and satisfaction scores between groups, and Pearson's correlation (r) will assess relationships between anxiety levels and satisfaction scores, while paired t-tests will be applied to compare anxiety levels before and after the intervention within groups. Additionally, multiple regression analysis will be employed to identify predictors of patient satisfaction and anxiety reduction, with a significance level set at p ≤ 0.05 for all statistical tests.Conclusion: The expected outcome of this study is that virtual reality-based education will significantly reduce pre-procedure anxiety and enhance patient satisfaction compared to standard education. Findings from this research may contribute to improving patient-centered care and developing innovative strategies to optimize emotional preparedness before cardiac catheterization procedures.

ELIGIBILITY:
Inclusion Criteria:

* • Adult patients (aged 18 years and above)

  * Scheduled for first-time elective cardiac catheterization
  * Able to understand Arabic or English
  * Capable of providing informed consent

Exclusion Criteria:

* • Individuals with cognitive impairment or psychiatric conditions that may interfere with their ability to engage in the VR intervention

  * Patients requiring emergency or urgent catheterization

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-03-05 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in pre-procedural anxiety (measured by DASS-21 Anxiety Subscale) | Baseline (before intervention) to immediately prior to cardiac catheterization (within 24 hours).
  Anxiety will be assessed using the Depression, Anxiety and Stress Scale - 21 (DASS-21). The Anxiety subscale includes 7 items, each scored 0-3. Subscale scores are multiplied by 2, giving a final range of 0-42. Higher scores indicate greater anxiety.